CLINICAL TRIAL: NCT05387980
Title: Special Investigation for CIBINQO （Long Term）
Brief Title: A Study to Learn About the Study Medicine (CIBINQO) in People With Atopic Dermatitis.
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7451055
Record Dates: First submitted 2022-05-09; First posted 2022-05-24 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis
Keywords: JAK Inhibitor; Atopic Dermatitis (AD); Abrocitinib; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients receiving CIBINQO: Patients receiving CIBINQO tablets by mouth for the treatment of Atopic Dermatitis.
  Interventions: Drug: CIBINQO

INTERVENTIONS:
Drug: CIBINQO — Patients receiving CIBINQO tablets by mouth for the treatment of Atopic Dermatitis.

SUMMARY:
The purpose of this study is to learn about the safety and effectiveness (how well the study treatment works) of the study medicine (CIBINQO) for the potential treatment of atopic dermatitis in people under Japanese medical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Participants receiving this Product for treatment of AD.
2. Participants start receiving this Product (commercial product) for the first time and no earlier than the contract date of this Study, or Participants who continues to receive this drug after hospital transfer can be registered retrospectively.

Exclusion Criteria:

1. Participants previously enrolled in this Study at the same site.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adolescent participants diagnosed with atopic dermatitis in Japan.
Sampling Method: Probability Sample
Enrollment: 1128 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2028-08-02 (Estimated); Study Completion 2028-08-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with adverse drug reactions | 156 weeks
Number of Participants with Discontinuation of Treatment | 156 weeks

SECONDARY OUTCOMES:
Percentage of Participants Achieving Investigator's Global Assessment (IGA) Score | Baseline, 156 weeks
  IGA Scores: Clear (0) or Almost Clear (1) and a Reduction From Baseline of Greater Than or Equal to ( >=2) Points at Week X: Non-responder Imputation
Percentage of Participants with Change From Baseline in Eczema Area and Severity Index (EASI) | Baseline, 156 weeks
Percentage of Participants with Change From Baseline in Affected % Body Surface Area (BSA) | Baseline, 156 weeks
Percentage of Participants with Change From Baseline in Pruritus Assessment | Baseline, 156 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Local Country Office, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451055